CLINICAL TRIAL: NCT04160234
Title: Web-based Preoperative Risk Assessment in the Elderly: a Pilot-study
Brief Title: Preoperative Risk Assessment in the Elderly
Acronym: PrepTAB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Ana Kowark, Consultant, RWTH Aachen University
Other Study IDs: EK 342/19
Record Dates: First submitted 2019-11-08; First posted 2019-11-12 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Preoperative Risk Assessment
Keywords: elderly; surgery; preoperative risk

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly patient: Preoperative elderly patients, who are planned for a surgical intervention
  Interventions: Other: web-based questionnaires

INTERVENTIONS:
Other: web-based questionnaires — Patients will be asked to complete web-based questionnaires on a tablet computer

SUMMARY:
PrepTAB aims to determine whether elderly patients are able to complete 4 preoperative risk assessment questionnaires within a web-based survey.

DETAILED DESCRIPTION:
Elderly patients are the most rapidly increasing group among surgical admissions. They are prone to a higher risk, because of predisposing risk factors. A comprehensive preoperative risk assessment is recommended by the European Society of Anaesthesiologists guideline, but time-consuming and usually not performed at present. A telemedical approach would enable an out-of hospital risk assessment before hospital admission and provide important information without the need for additional in-hospital resources. The feasibility of the completion of a web-based questionnaire by elderly patients, within a controlled in-hospital setting is required, as a base for a telemedical approach.

ELIGIBILITY:
Inclusion Criteria:

* Legally competent patients
* Written informed consent
* Age ≥ 65, male, female, diverse
* Multimorbid patients (≥ 2 comorbidities (according to the Charlson Comorbidity Index)
* Major elective surgery (such as total abdominal hysterectomy, endoscopic resection of prostate, lumbar discectomy, thyroidectomy, total joint replacement, lung operations, colon resection, radical neck dissection etc.)

Exclusion Criteria:

* Blind or deaf patients
* Patient/ Proxy not able to use electronic devices e.g. computer, tablet or smart phone
* Non-fluency in local language
* Alcohol and/ or drugs abuse
* Ambulatory surgery
* Repeated surgery, with previous participation
* Patients with severe neurological or psychiatric disorder
* Refusal of study participation by the patient

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: A convenient sample of patients, meeting all inclusion and none exclusion criteria, will be enrolled in the study. The patients will be recruited from the anaesthesia ambulance in the University hospital RWTH Aachen, where they have an appointment with the anaesthetist before their planned surgery.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-11-22 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Completion rate | 1 day
  The completion rate of the total number of questions of the web-based questionnaires

SECONDARY OUTCOMES:
Frequency of patient's requests for help to the accompanying next of kin | 1 day
  The study team member, who is present during the study treatment, will assess the frequency of the patient's requests for help to the accompanying next of kin
Assessment of the kind of patient's requests for help to the accompanying next of kin | 1 day
  The study team member, who is present during the study treatment, will assess the kind of the patient's requests for help to the accompanying next of kin, divided into: technical request or request regarding the content of the web-based questions
Assessment of the kind of patient's requests for help to the study team member | 1 day
  The study team member, who is present during the study treatment, will assess the kind of the patient's requests for help to himself, divided into: technical request or request regarding the content of the web-based questions
Frequency of patient's requests for help to the study team member | 1 day
  The study team member, who is present during the study treatment, will assess the frequency of the patient's requests for help to him
Elapsed time for questionnaire completion | 1 day
  The survey software will automatically count the elapsed time for completion of the questionnaires. The time will start in the moment, when the patient accesses the website and it will end when he presses the finish button
Ranking of unanswered questions | 1 day
  We will analyse which questions where not answered by the most patients.
Patient satisfaction | 1 day
  Analysis of patient satisfaction about the web-based questionnaires. A paper-based satisfaction questionnaire is provided to the patient after the completion of the web-based survey. The satisfaction questionnaire will consist of a 5-point Likert scale. It will consist of the items: Strongly disagree; Disagree; Neither agree nor disagree; Agree; Strongly agree
Frequency of technical problems | 1 day
  The frequency of technical problems (i.e. internet connection, black screen etc.) will be assessed by the present study team member

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, University Hospital Aachen, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No